CLINICAL TRIAL: NCT06890416
Title: A PHASE 3, MULTICENTER, PARALLEL-GROUP, OPEN-LABEL STUDY TO EVALUATE THE SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF RESPIRATORY SYNCYTIAL VIRUS PREFUSION F SUBUNIT VACCINE WHEN COADMINISTERED WITH HERPES ZOSTER SUBUNIT VACCINE IN ADULTS ≥50 YEARS OF AGE
Brief Title: A Study to Evaluate the Safety and Immunogenicity of RSVpreF Coadministered With Herpes Zoster Vaccine in Adults
Acronym: PISSARRO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: C3671058; PISSARRO (Other: Alias Study Number)
Record Dates: First submitted 2025-03-17; First posted 2025-03-24 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Respiratory Syncytial Virus (RSV)
Keywords: RSV; Vaccine
MeSH Terms: interventions — abrysvo

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Coadministration Group (Other): * Visit 1 (Day 1): RSVpreF + HZ/su dose 1
  * Visit 3 (Month 2): HZ/su dose 2
  Interventions: Biological: RESPIRATORY SYNCYTIAL VIRUS PREFUSION F SUBUNIT VACCINE; Biological: HZ/su VACCINE
- Sequential Administration Group (Other): * Visit 1 (Day 1): HZ/su dose 1
  * Visit 2 (Month 1): RSVpreF
  * Visit 3 (Month 2): HZ/su dose 2
  Interventions: Biological: RESPIRATORY SYNCYTIAL VIRUS PREFUSION F SUBUNIT VACCINE; Biological: HZ/su VACCINE

INTERVENTIONS:
Biological: RESPIRATORY SYNCYTIAL VIRUS PREFUSION F SUBUNIT VACCINE — Intramuscular injection
  Other Names: ABRYSVO; RSVpreF; PF-06928316
Biological: HZ/su VACCINE — intramuscular injection
  Other Names: SHINGRIX; RZV; HZ/su

SUMMARY:
This purpose of this phase 3 multicenter, parallel-group, open-label study is to learn about the safety, tolerability, and immunogenicity of RSVpreF and HZ/su vaccine when given together in adults 50 years of age and older.

ELIGIBILITY:
Inclusion Criteria

• Male and female participants 50 years of age and older who are healthy or with stable chronic medical conditions

Exclusion Criteria

* Current clinically suspected or polymerase chain reaction (PCR)-confirmed ongoing episode of HZ and/or history of clinically suspected or PCR-confirmed HZ within the past 12 months.
* Prior history of any subtype of Guillain Barré syndrome of any etiology.
* Serious chronic disorder, including metastatic malignancy, end-stage renal disease with or without dialysis, clinically unstable cardiac disease, or any other disorder that, in the investigator's opinion, excludes the participant from participating in the study.
* Immunocompromised individuals with known or suspected immunodeficiency, as determined by history and/or laboratory/physical examination, and medication list
* Previous vaccination with any licensed or investigational RSV vaccine at any time prior to enrollment, or planned receipt of a nonstudy RSV vaccine during study participation.
* Previous vaccination with any licensed recombinant adjuvant zoster vaccine (Shingrix) at any time prior to enrollment, or planned receipt of a nonstudy licensed VZV vaccine (Shingrix) during study participation.
* History of previous vaccination with live HZ vaccine (Zostavax) in the last 2 years from enrollment, or planned receipt through study participation.
* Previous vaccination with any investigational VZV vaccine at any time prior to enrollment, or planned receipt of a nonstudy investigational VZV vaccine during study participation.
* Individuals who receive chronic systemic treatment with immunosuppressive therapy, including cytotoxic agents, immunosuppressive monoclonal antibodies, systemic corticosteroids (defined as ≥20 mg/day of prednisone or equivalent for ≥14 days), eg, for cancer or an autoimmune disease, or radiotherapy, from 60 days before study intervention administration, or planned receipt throughout the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 526 (Actual)
Dates: Start 2025-04-04 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Geometric Mean Ratio (GMR) of Neutralizing Titer (NTs) for RSV A and B in RSVpreF + herpes zoster subunit vaccine (HZ/su) Compared to RSVpreF Alone | 1 month after vaccination with RSVpreF in the RSVpreF + HZ/su coadministration group to RSVpreF alone in the sequential administration group
Anti-gE antibody concentrations expressed as Geometric Mean Concentration (GMC) ratios in RSVpreF + HZ/su Compared to HZ/su Alone | 1 month after the second dose of HZ/su in the RSVpreF + HZ/su coadministration group to HZ/su alone in the sequential administration group
Percentage of Participants reporting Local Reactions Within 7 Days after Vaccination | Within 7 Days after each vaccination (Vaccination on Day 1)
  Describe local reactions (redness, swelling, and pain at the injection site) within 7 days following each study intervention administration recorded by participants in an electronic diary (e-diary).
Percentage of Participants with Systemic Events Within 7 Days after Vaccination | Within 7 Days after each vaccination (Vaccination on Day 1)
  Describe systemic events (fatigue, headache, vomiting, nausea, diarrhea, muscle pain, and joint pain) within 7 days following each study intervention administration recorded by participants in an electronic diary (e-diary).
Percentage of Participants with Adverse Events (AEs)from Vaccination through 1 Month after Vaccination | Within 1 Month after last vaccination
  Describe AEs occurring through 1 month after each study intervention administration
Percentage of Participants with Serious Adverse Events (SAEs) Throughout the Study | Within 4 Months after first study vaccination (Vaccination on Day 1)
  Describe SAEs occurring through 4 months after the first study intervention administration.

SECONDARY OUTCOMES:
NTs for RSV A and RSV B expressed as Geometric Mean Titers (GMT) | Before vaccination with RSVpreF, 1 month after vaccination with RSVpreF
NTs for RSV A and RSV B expressed as Geometric Mean Fold Rise (GMFR) | Before vaccination and 1 month after vaccination with RSVpreF
NTs for RSV A and RSV B expressed as seroresponse rate | 1 month after vaccination with RSVpreF
Anti-gE antibody concentrations expressed as GMCs | Before vaccination and 1 month after the second dose of HZ/su
Anti-gE antibody concentrations expressed as GMFRs | Before vaccination and 1 month after the second dose of HZ/su
Anti-gE antibody concentrations expressed as seroresponse rate | 1 month after the second dose of HZ/su

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (26):
- United States (25):
  - Central Research Associates, Birmingham, Alabama
  - Medical Affiliated Research Center, Huntsville, Alabama
  - AMR Clinical, Mobile, Alabama
  - Kaiser Permanente, Los Angeles, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Alliance for Multispecialty Research, LLC, Doral, Florida
  - Proactive Clinical Research,LLC, Fort Lauderdale, Florida
  - De La Cruz Research Center, LLC, Miami, Florida
  - Centricity Research Columbus Georgia Multispecialty, Columbus, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Synexus Clinical Research US, Inc., Chicago, Illinois
  - Optimal Research, Peoria, Illinois
  - DelRicht Research, New Orleans, Louisiana
  - Jadestone Clinical Research, Silver Spring, Maryland
  - Oakland Medical Research, Troy, Michigan
  - Clinical Research Professionals, Chesterfield, Missouri
  - IMA Clinical Research Warren, Warren Township, New Jersey
  - NYU Langone Health, New York, New York
  - Centricity Research Columbus Ohio Multispecialty, Columbus, Ohio
  - DM Clinical Research - Philadelphia, Philadelphia, Pennsylvania
  - Clinical Neuroscience Solutions Inc., Memphis, Tennessee
  - DM Clinical Research - Bellaire, Houston, Texas
  - SMS Clinical Research, Mesquite, Texas
  - IMA Clinical Research San Antonio, San Antonio, Texas
  - DM Clinical Research - Sugar Land, Sugar Land, Texas
- Clinical Research Puerto Rico, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3671058